CLINICAL TRIAL: NCT06981910
Title: The Effect of Psychoeducation on Body Image and Sexual Quality of Life in Patients Undergoing Mastectomy
Brief Title: The Role of Psychoeducation in Breast Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Çiçek SARUHAN, Lecturer, Dicle University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DicleU-ASBF-NURSE-ÇS-02
Record Dates: First submitted 2025-05-10; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Psychoeducation for Patients Who Have Undergone Mastectomy; Mastectomy
Keywords: Breast cancer; Mastectomy; Psychoeducation; Body image; Sexual quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study was carried out as a two-group, parallel, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation (Experimental): A semi-structured "Psychoeducation Program" was implemented over six weeks, with 90-minute sessions conducted weekly. Each subgroup received psychoeducation on different days within the same week. The week the psychoeducation concluded was designated as Week 0, and the scales were re-administered in Week 4.
  Interventions: Behavioral: Psychoeducation program
- Control (No Intervention): No intervention was provided to the control group; the same scales were administered to them during the 4th week after the conclusion of the psychoeducation program in the psychoeducation group

INTERVENTIONS:
Behavioral: Psychoeducation program — Each psychoeducation session included informational components, a preliminary group discussion of the topic, structured education on the discussed topic, awareness-raising activities within the group, opportunities for sharing, and emotional support. When participants' attention waned during sessions, breathing exercises were introduced. Depending on the group's preference, sessions concluded with a 2-3-minute poetry listening session and/or breathing exercises. At the end of each session, educational booklets prepared specifically for that session were distributed to the participants.
  Arms: Psychoeducation

SUMMARY:
This study aims to examine the effect of psychoeducation on body image and sexual quality of life in female patients who underwent mastectomy due to breast cancer.

DETAILED DESCRIPTION:
Method: This randomized controlled trial with two parallel groups was conducted between October 2023 and January 2025 in the general surgery clinic of a university hospital. The sample consisted of 63 patients (31 in the psychoeducation group and 32 in the control group). Data collection was conducted using the Patient Information Form, the Breast Cancer Body Image Scale (BCBIS), and the Sexual Quality of Life-Female (SQoL-F) questionnaire. Following the pretest administered to all participants, patients in the psychoeducation group received a 6-week psychoeducation program (90 minutes per week). After the completion of the 6-week intervention, a 4-week waiting period was implemented, after which the posttest was administered to all participants. Data analysis included descriptive statistics, chi-square test, t-test, Kolmogorov-Smirnov test, Cronbach's alpha coefficient, ANOVA, and Bonferroni post hoc tests.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 60 years
* Married and/or with a partner,
* Residing in the city where this study was carried out,
* İnformed about their diagnosis,
* With no physical deformities or functional impairments caused by comorbid conditions or treatments (e.g., lymphedema, hemiparesis, amputation, tracheostomy),
* Capable of communication, no cognitive impairments or diagnosed psychiatric disorders,
* Having completed chemotherapy and/or radiotherapy,
* With no prior counseling or education related to body image or sexual quality of life.

Exclusion Criteria:

* Women who were not between the ages of 18 and 60,
* Not married and/or without a partner,
* Not residing in the city where the study was conducted,
* Not informed about their diagnosis,
* With physical deformities or functional impairments caused by comorbid conditions or treatments (e.g., lymphedema, hemiparesis, amputation, tracheostomy),
* Unable to communicate, with cognitive impairments or diagnosed psychiatric disorders,
* Still undergoing chemotherapy and/or radiotherapy,
* Had previously received any counseling or education related to body image or sexual quality of life.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 63 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Body Image Scale (BCBIS) | 12 weeks
  The scale comprises 43 items (32 positively worded and 11 negatively worded) divided into two sections. Section 1 uses a five-point Likert scale: "Strongly disagree" (1), "Disagree" (2), "Neutral" (3), "Agree" (4), and "Strongly agree" (5). Section 2 also employs a five-point Likert scale: "Never" (1), "Rarely" (2), "Sometimes" (3), "Usually" (4), and "Always" (5). Negatively worded items are reverse-scored. The total score ranges between 43 and 215, and there is no established cutoff point; higher scores indicate a higher level of body image disturbance. The scale consists of six subdimensions. The Cronbach's α for the overall scale was reported to be 0.67.
Female Sexual Life Quality Scale (SQoL-F) | 12 weeks
  This 18-item scale has a six-point Likert format and was designed to be self-administered by women aged 18 and older. Participants are instructed to respond based on their sexual experiences during the past four weeks. Items are scored as follows: "Completely agree" (1), "Mostly agree" (2), "Somewhat agree" (3), "Somewhat disagree" (4), "Mostly disagree" (5), and "Completely disagree" (6). Before computing the total score (ranging from 18 to 108), responses to items 1, 5, 9, 13, and 18 are reverse-scored. The final score is converted to a scale out of 100, and a higher score indicates better sexual quality of life. The Cronbach's α for the overall scale is 0.83.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Özkan, Prof., Study Director — Department of Surgical Nursing, Faculty of Nursing, İnönü University
Locations (1):
- Dicle University Hospital, Diyarbakır, Turkey, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No